CLINICAL TRIAL: NCT05905068
Title: A Phase 1, Randomized, Single-blinded, Placebo-controlled, Single-ascending-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects of RN0191 in Adult Subjects With Elevated Low-Density Lipoprotein-Cholesterol
Brief Title: Adult Subjects With Elevated Low-Density Lipoprotein-Cholesterol to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ikaria Bioscience Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RN0191-101
Record Dates: First submitted 2023-06-02; First posted 2023-06-15 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: To Reduce the LDL-C Level in Hypercholesteremia Adult Patients; Combination for Subgroup High LDL-c Patients With Other Comorbidities

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo-controlled, single ascending-dose (SAD) study of RN0191 administered SC to adult subjects with elevated low-density lipoprotein-cholesterol. Subjects who have signed an Ethics Committee (EC)-approved informed consent form (ICF) and have met all the protocol eligibility criteria during screening may be enrolled into the study. In this SAD study, adult subjects with elevated LDL-C will be enrolled in up to 4 cohorts. Each cohort will comprise 8 subjects randomized in a 3:1 ratio (1:1 ratio for sentinel subjects; 5:1 ratio for non-sentinel subjects) to receive a single dose of RN0191 (n=6) or placebo (n=2), respectively.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 will be 25 mg RN0191 (or placebo) (Active Comparator)
  Interventions: Drug: RN0191 INJECTION
- Cohort 1 will be 100 mg RN0191 (or placebo) (Active Comparator)
  Interventions: Drug: RN0191 INJECTION
- Cohort 1 will be 300 mg RN0191 (or placebo) (Active Comparator)
  Interventions: Drug: RN0191 INJECTION
- Cohort 1 will be 500 mg RN0191 (or placebo) (Active Comparator)
  Interventions: Drug: RN0191 INJECTION

INTERVENTIONS:
Drug: RN0191 INJECTION — a sterile solution in each bottle for subcutaneous (SC) injection

SUMMARY:
Objectives: The primary and secondary objectives of the study are presented below. Exploratory objectives are presented in the body of the protocol.

Primary:

• To determine the safety and tolerability of RN0191 administered as escalating single subcutaneously (SC) doses in adult subjects with elevated low-density lipoprotein-cholesterol

Secondary:

* To evaluate the single-dose pharmacokinetics (PK) of RN0191 in adult subjects with elevated low-density lipoprotein-cholesterol
* To evaluate the pharmacodynamic (PD) effect of RN0191 on serum levels of low-density lipoprotein-cholesterol (LDL-C)
* To evaluate the PD effect of RN0191 on plasma levels of proprotein convertase subtilisin/kexin type 9 (PCSK9)

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, single ascending-dose (SAD) study of RN0191 administered SC to adult subjects with elevated low-density lipoprotein-cholesterol. Subjects who have signed an Ethics Committee (EC)-approved informed consent form (ICF) and have met all the protocol eligibility criteria during screening may be enrolled into the study. The study only has one part: SAD cohorts with Sentinel Dosing

The starting dose for subjects in Cohort 1 will be 25 mg RN0191 (or placebo). The following are the planned dose levels for subsequent cohorts in the SAD phase:

* Cohort 2: 100 mg RN0191 or placebo
* Cohort 3: 300 mg RN0191 or placebo
* Cohort 4: 500 mg RN0191 or placebo

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, aged 18 to 60 years, inclusive.
2. Body mass index between 18 and 32 kg/m2, inclusive, with body weight > 45 kg for females and >50 kg for males.
3. Serum LDL-C ≥100mg/dL (2.6 mmol/L) at screening and Day -1.
4. Fasting triglycerides < 400 mg/dL (<4.52 mmol/L) at screening and Day -1.
5. Adequate complete blood counts (complete blood counts [CBCs]; if outside the reference range, CBC values that are not clinically relevant and are acceptable to the Investigator)
6. Female subjects are eligible to participate if they are confirmed either not women of child-bearing potential (WOCBP), or have a negative urine pregnancy test at Day 1, are not breastfeeding, and willing and able to abide by the contraception guidelines.
7. Male subjects who can produce viable sperm are eligible to participate if they agree to use an adequate method of contraception as per the contraceptive guidance from Screening (signing the ICF) until at least 3 months post dose. Subjects with a partner(s) who is (are) not of childbearing potential are exempt from these requirements.
8. Male subjects with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile penetration. In addition, male subjects must refrain from donating sperm from Screening (signing the ICF) until at least 3 months post dose.
9. Willing to comply with protocol required visit schedule and visit requirements and provide written informed consent

Exclusion Criteria:

1. Male and female subjects, aged 18 to 60 years, inclusive.
2. Body mass index between 18 and 32 kg/m2, inclusive, with body weight > 45 kg for females and >50 kg for males .
3. Serum LDL-C ≥100mg/dL (2.6 mmol/L) at screening and Day -1.
4. Fasting triglycerides < 400 mg/dL (<4.52 mmol/L) at screening and Day -1.
5. Adequate complete blood counts (complete blood counts [CBCs]; if outside the reference range, CBC values that are not clinically relevant and are acceptable to the Investigator).
6. Female subjects are eligible to participate if they are confirmed either not women of child-bearing potential (WOCBP), or have a negative urine pregnancy test at Day 1, are not breastfeeding, and willing and able to abide by the contraception guidelines (signing the ICF).
7. Male subjects who can produce viable sperm are eligible to participate if they agree to use an adequate method of contraception as per the contraceptive guidance in Appendix 3 from Screening (signing the ICF) until at least 3 months post dose. Subjects with a partner(s) who is (are) not of childbearing potential are exempt from these requirements.
8. Male subjects with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile penetration. In addition, male subjects must refrain from donating sperm from Screening (signing the ICF) until at least 3 months post dose.
9. Willing to comply with protocol required visit schedule and visit requirements and provide written informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-02-24 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Exploratory objectives are presented in the body of the protocol. | For each subject in the study, the duration of the study clinic visits is approximately 21 weeks from screening to Day 85/EOS examination.
  • To determine the safety and tolerability of RN0191 administered as escalating single subcutaneously (SC) doses in adult subjects with elevated low-density lipoprotein-cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Kristi McLendon, MD, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Networks, Herston, Brisbane, Australia

IPD SHARING:
Plan to Share IPD: No